CLINICAL TRIAL: NCT05741424
Title: Single-center, Before-and-after Study Evaluating the Impact of BacT/Alert® VIRTUO®, BioFire® Blood Culture Identification 2-BCID2 and REVEAL® (bioMérieux) on the Optimization of Antibiotic Therapy for Gram-negative Bacteremia in the ICU Patient
Brief Title: Impact of BacT/Alert® VIRTUO®, BioFire® Blood Culture Identification 2-BCID2 and REVEAL® (bioMérieux) on the Optimization of Antibiotic Therapy for Gram-negative Bacteremia in the ICU
Acronym: BacteREVEAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Collaborators: BioMérieux (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: CIVI/2022/AP-01
Record Dates: First submitted 2023-02-14; First posted 2023-02-23 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Bacteremia
MeSH Terms: conditions — Bacteremia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- After innovative diagnostic technologies (Experimental)
  Interventions: Diagnostic Test: Innovative diagnostic technologies; Diagnostic Test: Reference diagnostic technique

INTERVENTIONS:
Diagnostic Test: Innovative diagnostic technologies — Samples from patients positive for Gram-negative bacteremia will be analyzed using the new BacT/Alert® VIRTUO®, BioFire® BCID2 and REVEAL® diagnostic solutions
Diagnostic Test: Reference diagnostic technique — Analysis of samples using diffusion on Mueller Hinton (MH) agar medium according to EUCAST.

SUMMARY:
Bacteremia is a frequent infection in intensive care units. It is associated with a high mortality rate and the rapid implementation of appropriate antibiotic therapy is strongly correlated to patient clinical outcomes.

Innovative technologies have emerged to shorten the turnaround time of blood culture samples by obtaining susceptibility testing of the incriminated pathogen at an early stage, and therefore to rapidly adjust the antibiotic therapy of patients with Gram-negative Bacilli bacteremia.

The study investigators hypothesize that the implementation of the innovative BacT/Alert® VIRTUO®, BioFire® BCID2 and REVEAL® solutions for the analysis of blood culture samples will increase the proportion of patients with Gram-negative Bacilli bacteremia who receive appropriate and optimized antibiotic therapy 24 hours after blood culture collection.

ELIGIBILITY:
Inclusion Criteria:

* The patient must be a member or beneficiary of a health insurance plan
* Patient admitted to the ICU with at least one positive blood culture for Gram-negative bacteremia

For the 'after' section of the study only:

* Patient must have given their free and informed consent or included by emergency procedure
* Patient signed the consent form or included by emergency procedure

Exclusion Criteria:

* The subject is participating in this study, or is in a period of exclusion determined by a previous study
* Consent refusal
* Patient with a polymicrobial blood culture
* Patient with a second episode of bacteremia
* Moribund patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-03-08 (Actual); Primary Completion 2024-05-06 (Actual); Study Completion 2024-06-16 (Actual)

PRIMARY OUTCOMES:
Proportion of patients receiving optimized antibiotic therapy (adequate and narrowest spectrum antibiotic therapy) in patients with Gram-negative bacteremia 24 hours after blood culture samples | 24 hours
  Yes/no: receiving optimized antibiotic therapy (effective and narrowest spectrum for the identified pathogen(s)) 24 hours after blood culture collection, before and after implementation of the new diagnostic solutions

SECONDARY OUTCOMES:
Time to adapt antibiotic therapy (optimized) based on susceptibility testing between the two periods of the study (before and after the implementation of innovative diagnostic technologies) following the collection of blood cultures | 28 Days
  Hours (theoretical and real) between blood culture collection and the first change in antibiotic therapy based on the innovative diagnostic technologies solutions or the conventional susceptibility test
Concordance of the REVEAL® rapid antibiotic susceptibility testing technology with reference methods | 28 Days
  Categorical Agreement of antibiotics tested by REVEAL® technology compared to the reference method (agar plate susceptibility test)
Patient survival | 28 Days
  Vital status of patients
Length of stay in intensive care unit | 28 Days
  Number of days
Prevalence rate of multiresistant bacteria between the "before" and "after" periods | 28 Days
  Proportion of multiresistant bacteria in each evaluation period
Prevalence rate of bacteria which are highly resistant to emerging antibiotics between the "before" and "after" periods | 28 Days
  Proportion of bacteria which are highly resistant to emerging antibiotics in each evaluation period
cost of the device for the healthcare facility | 28 Days
  purchase price of the equipment, depreciation, consumables, additional human time if applicable
Compare the amount per patient from the health insurance point of view. | 28 Days
  amount associated with the number of days spent in intensive care

CONTACTS AND LOCATIONS:
Overall Officials: Alix Pantel, Principal Investigator — CHU de Nimes; Claire Roger, Principal Investigator — CHU de Nimes
Locations (1):
- CHU de Nîmes, Nîmes, France

REFERENCES:
- [Result] Oudiane L, Benyahia M, Salipante F, Dubois A, Muller L, Lavigne JP, Pantel A, Roger C. Clinical impact of the BCID2 and rapid AST VITEK(R) REVEALTM on antibiotic optimisation in critically ill patients with Gram-negative bloodstream infections: a quasi-experimental pre/post interventional study. J Antimicrob Chemother. 2025 Oct 3;80(10):2665-2675. doi: 10.1093/jac/dkaf271. PMID 40754712